CLINICAL TRIAL: NCT03964155
Title: Assessment of a Novel Method for Non-invasive Sampling of the Distal Airspace in Acute Respiratory Distress Syndrome Patients Receiving Inhaled Sedation With Sevoflurane)
Brief Title: Sampling in ARDS Patients Under Inhaled Sedation
Acronym: ANAISS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical issues
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 JABAUDON 2 - ANAISS; 2018-A02596-49 (Other: ANSM)
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Acute Distress Respiratory
Keywords: Acute Respiratory Distress Syndrome; Inhaled Sedation with Sevoflurane; Biological collection
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Analysize correlation between sample from undiluted pulmonary edema andsample from AnaConDa-S® filter from patients presenting ARDS since 24 hours and sedated with inhaled sevoflurane.
Masking Description: The investigators and personals in charge of measuring protein markers in this study will be unaware of the fluid type (either AnaConDa-S® fluid,or undiluted pulmonary edema fluid or plasma). In addition, the study statistician will also be blinded during statistical analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with SDRA (Experimental): Patients within 24 hours from meeting the Berlin criteria for moderate or severe ARDS and receiving inhaled sedation with sevoflurane
  Interventions: Biological: Sample

INTERVENTIONS:
Biological: Sample — After an exposure duration of at least 12 hours, a sample of directly-aspirated, undiluted pulmonary edema fluid will be collected concurrently with AnaConDa-S® filter collection.

SUMMARY:
The main objective of this study is to compare the protein composition of simultaneously collected undiluted pulmonary edema fluid and AnaConDa-S ® fluid from patients with ARDS.

In a previous pilot randomized controlled trial, in patients with moderate-severe acute respiratory distress syndrome (ARDS), the use of inhaled sevoflurane improved oxygenation and decreased levels of a marker of lung epithelial injury (soluble receptor for advanced glycation end-products, sRAGE) and of some inflammatory markers (interleukin (IL)-1β, IL-6, IL-8 and tumor necrosis factor (TNF)-α), compared to intravenous midazolam. These results reinforce those from previously published preclinical studies as they suggest a protective effect of sevoflurane from alveolar/systemic inflammation and from reduced epithelial injury and/or improved alveolar fluid clearance, as assessed by plasma soluble receptor for advanced glycation end-products (sRAGE). The results from available studies support the safe use of sevoflurane inhalation through dedicated device is well tolerated, with no major adverse effect, e.g. on renal function or respiratory mechanics, in critically ill patients admitted to the intensive care unit (ICU), including those with ARDS.

Because the investigators group frequently uses sevoflurane in patients with ARDS and are interested in developing further research on the effects of inhaled sedation in ARDS, the current study has been designed to verify whether the same concept could be applied to the filter the investigators use to vaporize sevoflurane in their ICUs.

DETAILED DESCRIPTION:
Patients with moderate-to-severe ARDS (within 24 hours of onset) and already receiving inhaled sevoflurane for sedation as a current practice in participating centers will be enrolled in this observational study.

After an exposure duration of at least 12 hours, a sample of directly-aspirated, undiluted pulmonary edema fluid will be collected concurrently with AnaConDa-S®filter collection. This sample will be the only specific intervention of this study.

Patient data prospectively collected from the medical record will include demographics, ARDS risk factor, chest x-ray, ventilator settings at the time of AnaConDa-S ® filter collection, hospital and ICU length of stay and hospital mortality. Murray's lung injury score and the Acute Physiology and Chronic Health Evaluation (APACHE) II score will be calculated from data already available in the medical record.

AnaConDa-S ® filters will transported to the laboratory on ice and centrifuged at 2,000 x g for 10 minutes to collect condensed fluid that will be subsequently aliquoted and stored at -80°C for further analysis. Undiluted pulmonary edema fluid will be centrifuged at 2,000 x g for 10 minutes. Supernatants will be aliquoted and stored at - 80°C. Levels of IL-1β, IL-6, IL-8, TNF-α, soluble TNF-receptor 1, angiopoietin-2, and sRAGE will be measured in duplicate in both types of fluid with Multiplex.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients within 24 hours from meeting the Berlin criteria for moderate or severe ARDS and receiving inhaled sedation with sevoflurane will be eligible for inclusion into the study.

Exclusion Criteria:

* Patients <18 years
* Lack of deferred informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparaison between levels of protein markers, measured IL-1β, IL-6, IL-8, TNF-α, soluble TNF-receptor 1, angiopoietin-2, and sRAGE, measured in undiluted pulmonary edema fluid and in AnaConDa-S ® fluid | Between 12 hours and 24 hours after the begining of Sevoflurane sedation
  After an exposure duration of at least 12 hours, and when clinically available, a sample of directly-aspirated, undiluted pulmonary edema fluid will be collected (in general, only few ml are collected) concurrently with AnaConDa-S® filter collection. The concordance between levels of markers measured from undiluted alveolar fluid and those measured from AnaConDa-S® fluid will be explored using Lin's concordance coefficient, correlation coefficient (Pearson or Spearman according to the statistical distribution) and Bland-Altman plot. Confidence intervals at 95% will be presented. To complete these analyses, the satisfactory agreement will be confirmed by Passing and Bablok regression in order to highlight non-systematic and non-proportional differences between the two methods (undiluted pulmonary edema fluid and AnaConDa-S® fluid).

SECONDARY OUTCOMES:
Comparisons of levels of protein markers measured in AnaConDa-S® fluid between patients with focal ARDS and those with nonfocal ARDS | Between 12 hours and 24 hours after the begining of Sevoflurane sedation
  The levels of protein markers measured in AnaConDa-S® fluid will be compared between patients with focal ARDS and those with nonfocal ARDS using the unpaired t test or the Mann-Whitney U test when appropriate
The correlation between levels of protein markers measured in AnaConDa-S® and the Radiographic Assessment of Lung Edema (RALE) score developed recently by Pr. Lorraine Ware's team at Vanderbilt University. | Between 12 hours and 24 hours after the begining of Sevoflurane sedation
  The relationships between the levels of protein markers measured in AnaConDa-S® and the Radiographic Assessment of Lung Edema (RALE) score will be studied using correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Jabaudon, Principal Investigator — CHU de Clermont-Ferrand
Locations (2):
- France (2):
  - CHU, Clermont-Ferrand
  - CHU, Reims